CLINICAL TRIAL: NCT00210808
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Flexible-dose Study to Assess the Safety and Efficacy of Topiramate in the Treatment of Moderate to Severe Binge-eating Disorder Associated With Obesity
Brief Title: A Study of the Effectiveness and Safety of Topiramate in the Treatment of Moderate to Severe Binge-eating Disorder Associated With Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004657
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Binge-Eating Disorder
Keywords: Binge-Eating Disorder; medication treatment; obesity; bingeing
MeSH Terms: conditions — Obesity; Binge-Eating Disorder | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of topiramate compared to placebo in reducing the number of binge days in patients with moderate to severe binge-eating disorder associated with obesity.

DETAILED DESCRIPTION:
Binge-Eating Disorder (BED) is characterized by recurrent binge eating without extreme behaviors to lose weight (e.g., self-induced vomiting, misuse of laxatives) resulting in marked distress, feelings of loss of control, and association with overweight or obesity. Treatment goals for binge-eating therapies include reducing the urge to binge, weight loss, and management of co-existing medical and psychological conditions. Currently, there are no approved medication treatments available for BED, however, studies have shown that treatment for BED (psychotherapy or the use of medications) may be effective at reducing the number of binges, while effects on weight have been variable. Topiramate has been approved for epilepsy in adults and children aged 2 years and above, and for the prevention of migraine in adults. This is a randomized, double-blind, flexible dose, parallel group study to determine if topiramate, a prescription medication approved by the Food & Drug Administration for the treatment of epilepsy and the prevention of migraine, administered at a dose of 400 mg per day or the subject's maximum tolerated dose, is safe and effective compared with placebo in patients with moderate to severe binge-eating disorder associated with obesity. Subjects will have an equal chance of receiving topiramate or placebo. The study hypothesis is that topiramate will be more effective than placebo in reducing the number of binge days per week in patients with moderate to severe binge-eating disorder associated with obesity and is generally well tolerated. Patients completing the 16-week double-blind phase of the trial are eligible to participate in the 12-week open-label phase of the study.

Topiramate tablets (25 and/or 100 mg) or placebo in increasing doses starting at 25 mg/day up to 400 mg/ day (or MTD) during first 8 wks, achieved dose maintained for additional 8 wks. If entering OL reduce DB medication while increasing dose of active topiramate to 400mg/day or MTD for addn 12 wks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of binge-eating disorder
* 3 or more binge days per week in the 2 weeks prior to baseline
* Obese (body mass index >=30 and <=50 kilograms per square meter)
* Uncomplicated/controlled Type II diabetes or hypertension are acceptable
* In generally good health
* If female capable of having children, using acceptable method of birth control

Exclusion Criteria:

* No current or past history of schizophrenia, other psychotic disorder, or bipolar disorder
* Significant depression that requires treatment with medication or therapy
* At risk to self or others
* No current or recent (within 3 months) diagnosis of abusing drugs or alcohol
* Initiation of formal psychiatric therapy in past 6 months for binge-eating disorder or any other psychiatric disorder
* Pregnant or breast-feeding
* No clinically significant medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2003-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The rate of change in the number of binge days per week from baseline at 16 weeks or final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] McElroy SL, Hudson JI, Capece JA, Beyers K, Fisher AC, Rosenthal NR; Topiramate Binge Eating Disorder Research Group. Topiramate for the treatment of binge eating disorder associated with obesity: a placebo-controlled study. Biol Psychiatry. 2007 May 1;61(9):1039-48. doi: 10.1016/j.biopsych.2006.08.008. Epub 2007 Jan 29. PMID 17258690
- See also: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Study to Assess the Safety and Efficacy of Topiramate in the Treatment of Moderate to Severe Binge-Eating Disorder Associated with Obesity — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=614&filename=CR004657_CSR.pdf